CLINICAL TRIAL: NCT03088150
Title: COLLISION Trial - Colorectal Liver Metastases: Surgery vs Thermal Ablation, a Phase III Single-blind Prospective Randomized Controlled Trial
Brief Title: COLLISION Trial - Colorectal Liver Metastases: Surgery vs Thermal Ablation
Acronym: COLLISION
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Amsterdam UMC, location VUmc (Other)
Collaborators: Medtronic - MITG (Industry)
Responsible Party: Principal Investigator, Dr. M.R. Meijerink, Dr, Amsterdam UMC, location VUmc
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NL58551.029.16
Record Dates: First submitted 2017-01-11; First posted 2017-03-23 (Actual); Last update posted 2022-12-20 (Actual); Status verified 2022-12

CONDITIONS: ColoRectal Cancer; Liver Metastasis Colon Cancer; Liver Metastases; Surgery
Keywords: Hepatic resection; Liver surgery; Thermal ablation; Radiofrequency ablation; Microwave ablation; RFA; MWA
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Transurethral Resection of Prostate; Radiofrequency Ablation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Surgical resection (Active Comparator): Patients included will undergo resection of hepatic metastases, allowing thermal ablation for additional unresectable lesions.
  Interventions: Procedure: Surgical resection
- Thermal ablation (Experimental): Patients included will undergo ultrasound guided thermal ablation of hepatic metastases, allowing resection for additional unablatable lesions.
  Interventions: Procedure: Thermal ablation

INTERVENTIONS:
Procedure: Thermal ablation — Patients will undergo either radiofrequency ablation (RFA) or microwave ablation (MWA).
  Other Names: Radiofrequency ablation; RFA; Microwave ablation; MWA
  Arms: Thermal ablation
Procedure: Surgical resection — In case of randomization to surgical resection, the surgeon will remove all target lesions as well as all additional unablatable lesions.
  Arms: Surgical resection

SUMMARY:
The primary objective is to prove non-inferiority of thermal ablation compared to hepatic resection in patients with at least one resectable and ablatable colorectal liver metastases (≤3cm) and no extrahepatic disease.

DETAILED DESCRIPTION:
Study design:

COLLISION is a single-blind prospective multi-center phase-III randomized controlled trial. We hypothesize that thermal ablation is non-inferior to surgery for the selected patient groups in terms of the primary objective (overall survival). The Cox proportional hazards model (1-sided; non-inferiority or superiority) is used for sample size calculations. Given the superior safety profile we consider a hazard ratio of 1.3 to represent the upper limit of non-inferiority (non-inferiority margin). An HR of 1.3 corresponds to a 56.5% chance of the ablated patients to die first ((P = HR/(1 + HR) = 1.3/(1 + 1.3) = 0.565 (56.5%)). With 3 years of patient accrual and five years of follow-up we will have reached 60% of events (death) in approximately 6.5 years (overall probability of event, pE =0.6). The calculated sample size therefore is 599 (NS).To account for a 10% drop-out ratio (NDO=69) prior to randomization and a 3% loss to follow-up (NLTFU=18) after randomization we need to include 687 patients (NI). A total number of 618 patients will be randomized (NR) into one of two arms: arm A will undergo surgical resection (n=309) and arm B thermal ablation (n=309) for appointed target lesions.

Study population:

Patients with ≥1 resectable and ablatable CRLM (≤3cm), no extrahepatic disease and a good performance status (WHO 0-2) are considered eligible. Supplementary resections for resectable lesions >3cm and thermal ablations for unresectable CRLM ≤3cm are allowed with a maximum number of CRLM of 10.

Intervention:

Eligible patients will be stratified into low-, intermediate- and high disease burden after assessment by an expert panel. The panel, consisting of at least two diagnostic radiologists, two interventional radiologists and two hepatobiliary and/or oncological surgeons, will appoint lesions that are resectable and ablatable as target lesions, resectable and unablatable lesions as unablatable lesions and ablatable but unresectable lesions as unresectable lesions. All unablatable lesions should be resectable and all unresectable lesions should be ≤3cm and ablatable.

With the exception of patients that are suitable for laparoscopic resection or percutaneous ablation (low disease burden), eligibility needs to be reconfirmed during the surgical procedure. Hereafter patients will be randomized to undergo surgical resection of the target lesions (allowing thermal ablation for additional unresectable lesions) or thermal ablation (allowing resection for additional unablatable lesions). For open procedures randomization will be performed shortly after surgical inspection and IOUS with the patient under general anaesthesia. Both the experimenter(s) and the participant will be unaware of the eventual treatment arm prior to the procedure; after the procedure the patient will remain unaware (single-blind).

Conferring to national guidelines follow-up will include imaging, laboratory tests including tumour markers (CEA) and clinical examination every 3 months for the first year and every 6 months hereafter. Follow-up cross-sectional imaging should include at least an abdominal ceCT or upper abdominal ceMRI at the given time-points. Participating centres are free to add 18F-FDG PET-CTs at specific time-points or to use alternating specific modalities, as long as the follow-up protocol is pre-approved by the trial coordinators and as long as follow-up imaging is identical for both treatment arms. Quality of life questionnaires will be assessed at baseline, every 3 months for the first year and every 6 months hereafter accordingly.

Patients with recurrences that are considered unsuitable for additional focal therapy will be re-referred to their medical oncologist to assess additional systemic chemotherapy. In the event of chemotherapeutic down-staging hereafter, focal therapy can be reconsidered.

ELIGIBILITY:
Most important inclusion criteria:

* At least one CRLM size ≤ 3 cm eligible for both surgical resection and thermal ablation (target lesions);
* Additional unresectable CRLM should be ≤ 3 cm and ablatable (unresectable lesions);
* Additional unablatable CRLM should be resectable (unablatable lesions);
* Maximum number of CRLM 10;
* Resectability and ablatability should be re-confirmed intra-operatively by US plus full exploration for hepatic, peritoneal and regional lymph node metastases;
* ASA 1-3.

Most important exclusion criteria:

* No target lesions suitable for both resection and ablation;
* Radical treatment unfeasible or unsafe (e.g. insufficient FLR);
* The presence of extrahepatic nodal or non-nodal metastases;
* Immunotherapy or chemotherapy ≤ 6 weeks prior to the procedure;
* Any surgical resection or focal ablative liver therapy for CRLM prior to inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 618 (Estimated)
Dates: Start 2017-07-13 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | 5 years
  Counting from the date of randomization to the date of death of the patient or to the last day of follow-up.

SECONDARY OUTCOMES:
Disease free survival | 5 years
  The time from focal therapy to the time of events.
Time to progression | 5 years
  The time from focal therapy to the time of events.

CONTACTS AND LOCATIONS:
Overall Officials: MR Meijerink, MD, PhD, Principal Investigator — VU University Medical Center, Amsterdam, NL
Locations (1):
- Amsterdam University Medical Center - location VUmc, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] van der Lei S, Puijk RS, Dijkstra M, Schulz HH, Vos DJW, De Vries JJJ, Scheffer HJ, Lissenberg-Witte BI, Aldrighetti L, Arntz M, Barentsz MW, Besselink MG, Bracke B, Bruijnen RCG, Buffart TE, Burgmans MC, Chapelle T, Coolsen MME, de Boer SW, de Cobelli F, de Jong K, de Wilt JHW, Diederik AL, Dooper AMC, Draaisma WA, Eker HH, Erdmann JI, Futterer JJ, Geboers B, Groot GMC, Hagendoorn J, Hartgrink HH, Horsthuis K, Hurks R, Jenniskens SFM, Kater M, Kazemier G, Kist JW, Klaase JM, Knapen RRMM, Kruimer JWH, Lamers ABGN, Leclercq WKG, Liefers GJ, Manusama ER, Meier MAJ, Melenhorst MCAM, Mieog JSD, Molenaar QI, Nielsen K, Nijkamp MW, Nieuwenhuijs VB, Nota IMGC, Op de Beeck B, Overduin CG, Patijn GA, Potters FH, Ratti F, Rietema FJ, Ruiter SJS, Schouten EAC, Schreurs WH, Serafino G, Sietses C, Slooter GD, Smits MLJ, Soykan EA, Spaargaren GJ, Stommel MWJ, Timmer FEF, van Baardewijk LJ, van Dam RM, van Delden OM, van den Bemd BAT, van den Bergh JE, van den Boezem PB, van der Leij C, van der Meer RW, van der Meijs BBM, van der Ploeg APT, van der Reijden JJ, van Duijvendijk P, van Erkel AR, van Geel AM, Van Heek NT, van Manen CJ, van Rijswijk CSP, van Waesberghe JHTM, Versteeg KS, Vink T, Zijlstra IAJ, Zonderhuis BM, Swijnenburg RJ, van den Tol MP, Meijerink MR. Thermal ablation versus surgical resection of small-size colorectal liver metastases (COLLISION): an international, randomised, controlled, phase 3 non-inferiority trial. Lancet Oncol. 2025 Feb;26(2):187-199. doi: 10.1016/S1470-2045(24)00660-0. Epub 2025 Jan 20. PMID 39848272
- [Derived] Puijk RS, Ruarus AH, Vroomen LGPH, van Tilborg AAJM, Scheffer HJ, Nielsen K, de Jong MC, de Vries JJJ, Zonderhuis BM, Eker HH, Kazemier G, Verheul H, van der Meijs BB, van Dam L, Sorgedrager N, Coupe VMH, van den Tol PMP, Meijerink MR; COLLISION Trial Group. Colorectal liver metastases: surgery versus thermal ablation (COLLISION) - a phase III single-blind prospective randomized controlled trial. BMC Cancer. 2018 Aug 15;18(1):821. doi: 10.1186/s12885-018-4716-8. PMID 30111304